CLINICAL TRIAL: NCT06161077
Title: Voice Quality Analysis of Patients With Laryngotracheal Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00420355
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Subglottic Tracheal Stenosis
Keywords: Tracheal Stenosis; Voice Quality
MeSH Terms: conditions — Idiopathic subglottic tracheal stenosis; Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Voice Biomarker Screening Too — The investigators will develop a screening tool using voice that can predict disease severity in idiopathic subglottic stenosis

SUMMARY:
The investigators previously demonstrated that voice changes are common in patients with Laryngotracheal Stenosis (LTS), and patients typically report an improvement in voice outcomes following endoscopic dilation. Recently, NIH based programs such as a Bridge to Artificial Intelligence (Bridge2AI) have highlighted the use of artificial intelligence to identify acoustic biomarkers of disease. Therefore, the investigators hypothesize that progression of LTS scar can be quantified using acoustic measurements and machine learning. The goal of this clinical trial is to remotely monitor patient voice quality in an effort to determine if regularly performed voice recordings can be used as a diagnostic tool in order to predict the need for dilation procedures. The investigators feel that successful use of remote voice recording technology with algorithmic analysis will improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of laryngotracheal stenosis
* Patient age 18 - 80 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* The patient must be able to comprehend and have signed the informed consent.
* The patient must have documentation of their date of laryngotracheal stenosis diagnosis and prior medical/surgical history.

Exclusion Criteria:

* Inability to use the app associated with the study.
* Comorbid laryngeal or glottic disease
* Concurrent neurological disease which may impact voice use (such as tremor, parkinsonism, laryngeal dystonia)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with idiopathic subglottic stenosis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Voice Quality in patients with idiopathic subglottic stenosis | Baseline, 14 days, monthly for 2 years
  To remotely assess voice quality of patients with idiopathic subglottic stenosis with VoiceLab automated voice analysis software both before and at regular intervals following dilation procedures

SECONDARY OUTCOMES:
Change in Peak Expiratory flow (L/min) in patients with Laryngotracheal Stenosis | Baseline, 14 days, monthly for 2 years
  Change in Peak Expiratory flow (L/min) in patients with Laryngotracheal Stenosis will be assessed.
Change in Clinical COPD Questionnaire Quality of Life Score | Baseline, 14 days, monthly for 2 years
  Clinical COPD Questionnaire Quality of Life Score range of 0-6, with higher score indicating worse outcome
Change in Eating Assessment Tool (EAT-10) Swallow Quality of Life Score | Baseline, 14 days, monthly for 2 years
  Eating Assessment Tool (EAT-10) Swallow Quality of Life Score range of 0-40, with higher score indicating worse outcome
Change in 12-Item Short Form (SF-12) Survey Global Quality of Life Score | Baseline, 14 days, monthly for 2 years
  12-Item Short Form (SF-12) Survey Global Quality of Life Score of 0-100, with lower score indicating worse outcome
Change in lumen surface area | 2 years or when surgical intervention is required if before 2 years
  CT Neck will be used to assess change in lumen surface area in millimeters squared

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hillel, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States